CLINICAL TRIAL: NCT02036645
Title: A Randomised, Double-Blind, Placebo Controlled, Single and Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MEDI1814 in Subjects With Mild to Moderate Alzheimer's Disease.
Brief Title: SAD/MAD Study to Assess Safety, Tolerability, PK & PD of MEDI1814 in Subjects With Mild-Moderate Alzheimer's Disease.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D4750C00001
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Mild-Moderate Alzheimer's Disease; Healthy Elderly
MeSH Terms: interventions — Injections, Intravenous; Injections, Subcutaneous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- MEDI1814 IV (Experimental): Upto 10 cohorts of subjects are planned to be dosed by IV injection, with single and multiple ascending doses ranging from 25-1800mg.
  Interventions: Biological: MEDI1814 for IV injection
- IV Placebo (Placebo Comparator): Upto 10 cohorts of subjects are planned to be dosed by IV injection, with single and multiple ascending doses ranging from 25-1800mg.
  Interventions: Biological: MEDI1814 for IV injection; Biological: IV Placebo
- MEDI1814 Sub Cutaneous Injection (Experimental): 2 cohorts of subjects are planned to be dosed by sub cutaneous injection, one single ascending dose and one multiple ascending dose cohort
  Interventions: Biological: MEDI1814 for Subcutaneous Injection
- Subcutaneous Placebo (Placebo Comparator): 2 cohorts of subjects are planned to be dosed by sub cutaneous injection, one single ascending dose and one multiple ascending dose cohort
  Interventions: Biological: Placebo for Subcutaneous Injection

INTERVENTIONS:
Biological: MEDI1814 for IV injection — Monoclonal antibody for IV Injection
  Arms: IV Placebo; MEDI1814 IV
Biological: MEDI1814 for Subcutaneous Injection — Monoclonal antibody for subcutaneous injection
  Arms: MEDI1814 Sub Cutaneous Injection
Biological: IV Placebo — Placebo for IV injection
  Arms: IV Placebo
Biological: Placebo for Subcutaneous Injection — Subcutaneous Placebo Injection
  Arms: Subcutaneous Placebo

SUMMARY:
The purpose of this study is to assess the safety, drug levels and effects on the body of 1 or 3 injections of MEDI1814, in people with mild to moderate Alzhiemer's Disease or healthy elderly people.

ELIGIBILITY:
Inclusion Criteria Male and female (non child bearing potential) subjects Mild-moderate Alzheimer's Disease

Exclusion Criteria History or evidence of significant autoimmune disease Presence of psychiatric disorder which would affect completion of the study Current serious or unstable clinically important illness

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-02-04 (Actual); Primary Completion 2016-09-15 (Actual); Study Completion 2016-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thor Ostenfeld, MD, Study Director — AstraZeneca; David Han, MD, Principal Investigator — Glendale Parexel Early Phase Clinical Unit
Locations (10):
- United States (10):
  - Research Site, Glendale, California
  - Research Site, Long Beach, California
  - Research Site, Panorama City, California
  - Research Site, Hallandale, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Baltimore, Maryland
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 261 screening visits in 193 individuals were required to randomize 45 subjects into 6 Single Ascending Dose (SAD) cohorts and 32 subjects into 4 Multiple Ascending Dose (MAD) cohorts.
Pre-assignment Details: Due to population (mild to moderate Alzheimer's disease) and duration (6 or 9 months) per cohort, rescreening was permitted. SAD had 128 screeings in105 subjects (23 rescreens); MAD had 133 screenings in 88 subjects, (22 rescreens from SAD and 23 rescreens from MAD). Note: 11 of 32 randomized MAD subjects had previously completed a SAD cohort.
Groups:
- Placebo: SAD: Placebo: pooled SAD pooled cohorts 1, 2, 3, 4, 5 IV & 6 SC (2 subjects each)
- Medi1814 25 mg IV: SAD: Medi1814 25 mg IV: SAD cohort 1
- Medi1814 100 mg IV: SAD: Medi1814 100 mg IV: SAD cohort 2
- Medi1814 300 mg IV: SAD: Medi1814 300 mg IV: SAD cohort 3
- Medi1814 900 mg IV: SAD: Medi1814 900 mg IV: SAD cohort 4
- Medi1814 1800 mg IV: SAD: Medi1814 1800 mg IV: SAD cohort 5
- Medi1814 100 mg SC: SAD: Medi1814 100 mg SC: CAD cohort 6
- Placebo: MAD: Placebo: MAD pooled cohorts 7, 8, 9 IV & 10 SC (2 subjects each)
- Medi1814 300 mg IV: MAD: Medi1814 300 mg IV: MAD cohort 7
- Medi1814 900 mg IV: MAD: Medi1814 900 mg IV: MAD cohort 8
- Medi1814 1800 mg IV: MAD: Medi1814 1800 mg IV: MAD cohort 9
- Medi1814 200 mg SC: MAD: Medi1814 200 mg SC: MAD cohort 10
Period: SAD Cohorts : Study Part 1
Arm/Group | Placebo: SAD | Medi1814 25 mg IV: SAD | Medi1814 100 mg IV: SAD | Medi1814 300 mg IV: SAD | Medi1814 900 mg IV: SAD | Medi1814 1800 mg IV: SAD | Medi1814 100 mg SC: SAD | Placebo: MAD | Medi1814 300 mg IV: MAD | Medi1814 900 mg IV: MAD | Medi1814 1800 mg IV: MAD | Medi1814 200 mg SC: MAD
Started | 12 (Pooled across cohorts 1-5 (2 per cohort)) | 3 | 6 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0
Completed | 12 | 3 | 6 | 5 | 6 | 6 | 5 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: MAD Cohorts: Study Part 2
Arm/Group | Placebo: SAD | Medi1814 25 mg IV: SAD | Medi1814 100 mg IV: SAD | Medi1814 300 mg IV: SAD | Medi1814 900 mg IV: SAD | Medi1814 1800 mg IV: SAD | Medi1814 100 mg SC: SAD | Placebo: MAD | Medi1814 300 mg IV: MAD | Medi1814 900 mg IV: MAD | Medi1814 1800 mg IV: MAD | Medi1814 200 mg SC: MAD
Started | 0 (Pooled across Cohorts 7 to 9 (2 per cohort)) | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 6 | 6 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized subjects, Safety Analysis Population
Groups:
- Medi 1814 900 mg IV: MAD: Medi1814 900 mg IV: MAD cohort 8
- Total: Total of all reporting groups
Arm/Group | Placebo: SAD | Medi1814 25 mg IV: SAD | Medi1814 100 mg IV: SAD | Medi1814 300 mg IV: SAD | Medi1814 900 mg IV: SAD | Medi1814 1800 mg IV: SAD | Medi1814 100 mg SC: SAD | Placebo: MAD | Medi1814 300 mg IV: MAD | Medi 1814 900 mg IV: MAD | Medi1814 1800 mg IV: MAD | Medi1814 200 mg SC: MAD | Total
Number analyzed (Participants) | 12 | 3 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (7.22) [55 to 79] | 74.0 (8.89) [67 to 84] | 66.8 (1.94) [64 to 69] | 69.0 (6.10) [59 to 77] | 71.8 (5.15) [66 to 78] | 64.8 (5.91) [56 to 73] | 69.3 (4.84) [65 to 78] | 70.0 (5.90) [63 to 80] | 71.7 (6.62) [65 to 80] | 70.8 (6.62) [55 to 70] | 62.5 (6.16) [56 to 79] | 69.3 (8.71) | 68.5 (6.55) [55 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 0 | 6 | 5 | 4 | 1 | 3 | 5 | 3 | 2 | 3 | 5 | 44
  Male | 5 | 3 | 0 | 1 | 2 | 5 | 3 | 3 | 3 | 4 | 3 | 1 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 0 | 5 | 4 | 1 | 6 | 1 | 5 | 5 | 5 | 6 | 6 | 52
  Not Hispanic or Latino | 4 | 3 | 1 | 2 | 5 | 0 | 5 | 3 | 1 | 1 | 0 | 0 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
  White | 10 | 1 | 6 | 4 | 5 | 6 | 5 | 8 | 5 | 6 | 6 | 5 | 67
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mini Mental State Exam (MMSE) [Mean (Standard Deviation); unit: MMSE score] — Mini Mental State Exam (MMSE) - indicator of dementia; range of score of enrolled subjects 16 to 26, Scale range 0 to 30, higher score worse
  MMSE score | 21.8 (3.02) | 22.0 (2.65) | 22.3 (3.27) | 22.5 (3.73) | 22.2 (2.99) | 21.0 (2.00) | 23.2 (2.04) | 22.1 (2.48) | 19.8 (2.58) | 20.2 (1.72) | 20.0 (2.45) | 22.5 (2.59) | 21.6 (3.07)

OUTCOME MEASURES:

1. Primary Outcome: Tolerability as Measured by Participant Withdrawal for an Adverse Event
Description: Tolerability measured by participant withdrawal for an adverse event from randomization through end of study
Time Frame: 4 months SAD; 7 months MAD
Population: Safety Population
Measure: Number; unit: Participants
Groups:
- Medi1814 100 mg SC : SAD: Medi1814 100 mg SC: SAD cohort 6
Arm/Group | Placebo: SAD | Medi1814 25 mg IV: SAD | Medi1814 100 mg IV: SAD | Medi1814 300 mg IV: SAD | Medi1814 900 mg IV: SAD | Medi1814 1800 mg IV: SAD | Medi1814 100 mg SC : SAD | Placebo: MAD | Medi1814 300 mg IV: MAD | Medi1814 900 mg IV: MAD | Medi1814 1800 mg IV: MAD | Medi1814 200 mg SC: MAD
Number analyzed (Participants) | 12 | 3 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Area Under the Concentration Time Curve (AUC) Time 0 to t (28 Days After 1st Dose SAD and MAD and After 3rd Dose in MAD, Day 57)
Description: Area Under the Concentration time curve (AUC) time 0 to t; calculated from Just prior to dose administration start to 28th day after dose (pre infusion, during infusion, 1,2,4,8,24,48 hr 7, 14, 21, and 28 day)
Time Frame: 1 month
Population: Pharmacokinetic Population (subjects treated with Medi1814)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng x day/mL
Arm/Group | Medi1814 25 mg IV: SAD | Medi1814 100 mg IV: SAD | Medi1814 300 mg IV: SAD | Medi1814 900 mg IV: SAD | Medi1814 1800 mg IV: SAD | Medi1814 100 mg SC: SAD | Medi1814 300 mg IV: MAD | Medi1814 900 mg IV: MAD | Medi1814 1800 mg IV: MAD | Medi1814 200 mg SC: MAD
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng x day/mL
  First Dose (day 1-29) | 80.5 (61.1) | 455 (19.7) | 1550 (26.3) | 4040 (28.0) | 4420 (30.7) | 120 (51.9) | 710 (24.2) | 1690 (75.3) | 4490 (24.2) | 162 (69.2)
  Third dose (day 57-85) | NA (NA) — single dose only | NA (NA) — single dose only | NA (NA) — single dose only | NA (NA) — single dose only | NA (NA) — single dose only | NA (NA) — single dose only | 1150 (37.9) | 2680 (74) | 7150 (27.3) | 134 (57.0)
Statistical Analysis 1: Comparison: Medi1814 25 mg IV: SAD vs Medi1814 100 mg IV: SAD vs Medi1814 300 mg IV: SAD vs Medi1814 900 mg IV: SAD vs Medi1814 1800 mg IV: SAD; Test type: Superiority or Other; Regression, Linear; Slope = 0.93, 95% CI 2-sided [0.82 to 1.04] — Since an Estimation approach was taken for the statistical analysis, no p-values were calculated
Statistical Analysis 2: Comparison: Medi1814 300 mg IV: MAD vs Medi1814 900 mg IV: MAD vs Medi1814 1800 mg IV: MAD; Test type: Superiority or Other; Regression, Linear; Slope = 1.01, 95% CI 2-sided [0.71 to 1.30] — Since an Estimation approach was taken for the statistical analysis, no p-values were calculated

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Medi1814
Description: Maximum plasma concentration (Cmax) of Medi1814 during 28 day period after dose administration start (prior to dosing, during infusion, 1, 2, 4, 8, 24, 48 hr, 7, 14,21, and 28 days)
Time Frame: 1 month
Population: Pharmacokinetic population (subjects dosed with Medi1814)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Medi1814 25 mg IV: SAD | Medi1814 100 mg IV: SAD | Medi1814 300 mg IV: SAD | Medi1814 900 mg IV: SAD | Medi1814 1800 mg IV: SAD | Medi1814 100 mg SC: SAD | Medi1814 300 mg IV: MAD | Medi1814 900 mg IV: MAD | Medi1814 1800 mg IV: MAD | Medi1814 200 mg SC: MAD
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng/ml
  First dose (day 1-29) | 10.2 (42.7) | 38.7 (30.9) | 102 (14.7) | 341 (19.3) | 424 (36.1) | 3.59 (51.4) | 83.9 (22.3) | 172 (77.2) | 496 (24.4) | 10.1 (81.4)
  Third dose (day 57-85) | NA (NA) — SAD - Day 1 dose only | NA (NA) — SAD - Day 1 dose only | NA (NA) — SAD - Day 1 dose only | NA (NA) — SAD - Day 1 dose only | NA (NA) — SAD - Day 1 dose only | NA (NA) — SAD - Day 1 dose only | 96.7 (38.3) | 185 (110) | 536 (32.3) | 7.56 (38.5)
Statistical Analysis 1: Comparison: Medi1814 25 mg IV: SAD vs Medi1814 100 mg IV: SAD vs Medi1814 300 mg IV: SAD vs Medi1814 900 mg IV: SAD vs Medi1814 1800 mg IV: SAD; Test type: Superiority or Other; Regression, Linear; Slope = 0.90, 95% CI 2-sided [0.81 to 0.98] — Since an Estimation approach was taken for the statistical analysis, no p-values were calculated
Statistical Analysis 2: Comparison: Medi1814 300 mg IV: MAD vs Medi1814 900 mg IV: MAD vs Medi1814 1800 mg IV: MAD; Test type: Superiority or Other; Regression, Linear; Slope = 0.96, 95% CI 2-sided [0.65 to 1.27] — Since an Estimation approach was taken for the statistical analysis, no p-values were calculated

4. Secondary Outcome: Mean Termination Half Life (t 1/2) of Medi1814
Description: Mean termination half life (t 1/2) of Medi1814 during 28 day period after dose administration start (SAD Day 1 dose, MAD 3rd dose)
Time Frame: 1 month
Population: Pharmacokinetic population (subjects dosed with Medi1814)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Medi1814 25 mg IV: SAD | Medi1814 100 mg IV: SAD | Medi1814 300 mg IV: SAD | Medi1814 900 mg IV: SAD | Medi1814 1800 mg IV: SAD | Medi1814 100 mg SC: SAD | Medi1814 300 mg IV: MAD | Medi1814 900 mg IV: MAD | Medi1814 1800 mg IV: MAD | Medi1814 200 mg SC: MAD
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
days
  First dose (day 1-29) | 17.2 (0.94) | 17.0 (2.16) | 17.1 (2.78) | 19.0 (2.23) | 18.3 (7.69) | 19.8 (3.56) | NA (NA) — MAD not assessed after 1st dose | NA (NA) — MAD not assessed after 1st dose | NA (NA) — MAD not assessed after 1st dose | NA (NA) — MAD not assessed after 1st dose
  Third dose (day 57-85) | NA (NA) — SAD had 1 dose only | NA (NA) — SAD had 1 dose only | NA (NA) — SAD had 1 dose only | NA (NA) — SAD had 1 dose only | NA (NA) — SAD had 1 dose only | NA (NA) — SAD had 1 dose only | 14.2 (1.86) | 16.2 (1.61) | 20.4 (5.38) | 16.4 (3.29)

5. Secondary Outcome: Biomarkers: Amyloid-beta in Cerebral Spinal Fluid (Two Amyloid Bets Peptides of 40 and 42 Amino Acids Were Assessed)
Description: Biomarkers: Amyloid-beta in cerebral spinal fluid, mean percent change from baseline
Time Frame: Day 29 in SAD; Day 85 in MAD
Population: Pharmacodynamic population (with non zero baseline values)
Measure: Mean (Standard Deviation); unit: % change
Groups:
- Medi1814 900 mg: MAD: Medi1814 900 mg IV: MAD cohort
Arm/Group | Placebo: SAD | Medi1814 25 mg IV: SAD | Medi1814 100 mg IV: SAD | Medi1814 300 mg IV: SAD | Medi1814 900 mg IV: SAD | Medi1814 1800 mg IV: SAD | Medi1814 100 mg SC: SAD | Placebo: MAD | Medi1814 300 mg IV: MAD | Medi1814 900 mg: MAD | Medi1814 1800 mg IV: MAD | Medi1814 200 mg SC: MAD
Number analyzed (Participants) | 12 | 3 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6
% change
  Total amyloid-beta 1-40 | 122.9 (426.51) | -15.9 (20.57) | -21.0 (19.57) | 8.72 (31.69) | 2.0 (29.21) | 10.2 (98.14) | -14.6 (23.69) | 4.96 (90.19) | 638.5 (1054.28) | -17.9 (34.08) | -36.96 (46.82) | 38.06 (47.51)
  Total amyloid-beta 1-42 | 25.3 (100.71) | 52.0 (104.35) | 41.7 (38.68) | 192.8 (127.96) | 414.7 (292.18) | 376.1 (295.92) | 5.87 (24.52) | -29.4 (55.90) | 633.6 (471.79) | 197.5 (115.25) | 915.5 (1361.86) | 87.8 (124.68)
  Free amyloid-beta 1-42 | 28.6 (113.70) | -33.9 (13.98) | -54.3 (39.96) | -57.2 (55.80) | -81.65 (21.67) | -15.2 (189.05) | -19.0 (17.69) | -2.5 (62.66) | 11.6 (167.59) | -96.3 (2.26) | -95.0 (1.88) | -57.7 (29.76)

6. Secondary Outcome: Biomarker: Total Amyloid-beta 1-42 in Plasma
Description: Biomarker: Total Amyloid-beta 1-42 in plasma, mean percent change from baseline
Time Frame: Day 29 in SAD; Day 85 in MAD
Population: Pharmacodynamic population (with non zero baseline values)
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Placebo: SAD | Medi1814 25 mg IV: SAD | Medi1814 100 mg IV: SAD | Medi1814 300 mg IV: SAD | Medi1814 900 mg IV: SAD | Medi1814 1800 mg IV: SAD | Medi1814 100 mg SC: SAD | Placebo: MAD | Medi1814 300 mg IV: MAD | Medi1814 900 mg IV: MAD | Medi1814 1800 mg IV: MAD | Medi1814 200 mg SC: MAD
Number analyzed (Participants) | 12 | 3 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6
% change | 19.6 (34.51) | 40132.5 (4379.93) | 41107.0 (43509.89) | 46667.9 (29628.09) | 78534.5 (22773.96) | 44050.9 (15776.40) | 45404.0 (1808.13) | -32.0 (45.65) | 30272.4 (14834.80) | 84652.8 (44649.16) | 43415.3 (13760.07) | 97140.1 (34151.47)

7. Secondary Outcome: Medi1814 Concentration in CSF Samples
Description: Medi1814 concentration in CSF Samples; number of sampled subjects with a value above the lower limit of quantification
Time Frame: SAD Day 29; MAD Day 85
Population: Pharmacokinetic population (subjects dosed with Medi1814)
Measure: Number; unit: Participants
Arm/Group | Medi1814 25 mg IV: SAD | Medi1814 100 mg IV: SAD | Medi1814 300 mg IV: SAD | Medi1814 900 mg IV: SAD | Medi1814 1800 mg IV: SAD | Medi1814 100 mg SC: SAD | Medi1814 300 mg IV: MAD | Medi1814 900 mg IV: MAD | Medi1814 1800 mg IV: MAD | Medi1814 200 mg SC: MAD
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  First dose (day 1-29) | 0 (0.94) | 0 (2.16) | 1 (2.78) | 2 (2.23) | 4 (7.69) | 0 (3.56) | NA (NA) — MAD not assessed after first dose | NA (NA) — MAD not assessed after first dose | NA (NA) — MAD not assessed after first dose | NA (NA) — MAD not assessed after first dose
  Third dose (day 57-85) | NA (NA) — SAD only 1 dose | NA (NA) — SAD only 1 dose | NA (NA) — SAD only 1 dose | NA (NA) — SAD only 1 dose | NA (NA) — SAD only 1 dose | NA (NA) — SAD only 1 dose | 1 (1.86) | 5 (1.61) | 6 (5.38) | 0 (3.29)

8. Secondary Outcome: Immunogenicity: Anti-drug Antibody Titer
Description: Immunogenicity: Anti-drug antibody titer, subject counted if titer 50 or greater on any test, else 0 if all <50
Time Frame: 4 months SAD (6 tests over 4 months; week 1, 2, 4, 8, 12, 16); 7 months MAD (7 monthly tests)
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo: SAD | Medi1814 25 mg IV: SAD | Medi1814 100 mg IV: SAD | Medi1814 300 mg IV: SAD | Medi1814 900 mg IV: SAD | Medi1814 1800 mg IV: SAD | Medi1814 100 mg SC : SAD | Placebo: MAD | Medi1814 300 mg IV: MAD | Medi1814 900 mg IV: MAD | Medi1814 1800 mg IV: MAD | Medi1814 200 mg SC: MAD
Number analyzed (Participants) | 12 | 3 | 6 | 6 | 6 | 6 | 6 | 8 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline until day 113 (4 months) in SAD Study Part 1; From baseline until day 169 (7 months) in MAD Study Part 2
Description: Treatment emergent from day of randomization until 4 months after the last dose administration (IV = intravenous dosing; SC = subcutaneous dosing)
Arm/Group | Placebo: SAD | Medi1814 25 mg IV: SAD | Medi1814 100 mg IV: SAD | Medi1814 300 mg IV: SAD | Medi1814 900 mg IV: SAD | Medi1814 1800 mg IV: SAD | Medi1814 100 mg SC: SAD | Placebo: MAD | Medi1814 300 mg IV: MAD | Medi1814 900 mg IV: MAD | Medi1814 1800 mg IV: MAD | Medi1814 200 mg SC: MAD
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/3 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/3 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 5/12 | 1/3 | 3/6 | 3/6 | 6/6 | 1/6 | 4/6 | 3/8 | 4/6 | 3/6 | 2/6 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo: SAD (N=12) | Medi1814 25 mg IV: SAD (N=3) | Medi1814 100 mg IV: SAD (N=6) | Medi1814 300 mg IV: SAD (N=6) | Medi1814 900 mg IV: SAD (N=6) | Medi1814 1800 mg IV: SAD (N=6) | Medi1814 100 mg SC: SAD (N=6) | Placebo: MAD (N=8) | Medi1814 300 mg IV: MAD (N=6) | Medi1814 900 mg IV: MAD (N=6) | Medi1814 1800 mg IV: MAD (N=6) | Medi1814 200 mg SC: MAD (N=6)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Occipital neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Although 11 subjects were in both a SAD and a MAD cohort, summaries were for those assigned to the cohort regardless of participation in any other cohort

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No